CLINICAL TRIAL: NCT00212381
Title: Diindolylmethane (DIM) Dietary Supplementation: A Nonsurgical Treatment for Cervical Intraepithelial Neoplasia (CIN)
Brief Title: Oral Diindolylmethane (DIM) for the Treatment of Cervical Dysplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Del Priore, Professor, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9218; NCT00206804 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Cervical Dysplasia
Keywords: cervical dysplasia, diindolylmethane, pap smear
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: randomized double blind intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: central pharmacy dispenses based on sealed randomization table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral DIM (Active agent) (Experimental): 2mg/kg/day po of DIM
  Interventions: Drug: di indolylmethane (DIM)
- Red rice bran (Placebo) (Active Comparator): this agent is not generally thought to be active but may be
  Interventions: Dietary Supplement: Red rice bran

INTERVENTIONS:
Drug: di indolylmethane (DIM) — This is the agent being studies. Similar agents have been reported to have potential activity.
  Arms: oral DIM (Active agent)
Dietary Supplement: Red rice bran — this will act as the active comparator. The sponsor provided this as the "placebo" arm since it is a filler component of their DIM capsules
  Arms: Red rice bran (Placebo)

SUMMARY:
To determine if the use of oral Diindolylmethante (DIM), a marketed cruciferous vegetable based dietary supplement (Bioresponse-DIM), is associated with the regression of cervical dysplasia in otherwise healthy women.

DETAILED DESCRIPTION:
To determine if the use of oral Diindolylmethane (DIM), a marketed cruciferous vegetable based dietary supplement (BioResponse-DIM®), is associated with the regression of cervical dysplasia in otherwise healthy women. Additionally, the study aims to see how the use of the BioResponse-DIM supplement correlates with cervical HPV colonization, and to asses the tolerability of daily DIM supplementation

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women greater than or equal to 18 years of age able to consent
* CIN II or III confirmed by histology
* Karnofsky performance status >= 80
* No prior treatment for dysplasia in the past 4 months

Exclusion Criteria:

* Incompletely visible lesion
* Diethylstilbestrol (DES) exposure
* HIV seropositive

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2000-09; Primary Completion 2006-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Measure the regression of CIN in women by cytology, colposcopy, and biopsy, | 3 months
  To determine if oral DIM is effective in promoting the regression of CIN in women

SECONDARY OUTCOMES:
HPV colonization by commercial ELIZA test | 3 months
  To correlate the response to DIM with HPV colonization
Adverse events reported by subjects and lab abnormalities i.e. CBC and SMA20 | one year
  To assess for any adverse effects of oral DIM in women

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Del Priore, M.D., M.P.H., Study Director — NY Downtown Hospital; Alan Arslan, M.D., Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Del Priore G, Gudipudi DK, Montemarano N, Restivo AM, Malanowska-Stega J, Arslan AA. Oral diindolylmethane (DIM): pilot evaluation of a nonsurgical treatment for cervical dysplasia. Gynecol Oncol. 2010 Mar;116(3):464-7. doi: 10.1016/j.ygyno.2009.10.060. Epub 2009 Nov 24. PMID 19939441